CLINICAL TRIAL: NCT06736977
Title: Effectiveness of Nurse-Led Education Programmes to Enhance Infection Prevention and Control Among Childcare Workers in Bangkok Daycare Centres, Thailand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Chakkrich Pidjadee, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: COA.1-051/2024
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Hand Hygiene Behavior; Infection Control; Infection Prevention
Keywords: Nurse-led education programme; Infection control; Knowledge; Attitude; Practice; Self-efficacy; Hand hygiene intention; Hand hygiene compliance; Childcare worker; Child day care centres
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The Onsite Nurse-Led Education Programme on IPC (Experimental): The researcher will conduct the Nurse-Led Education Programme on IPC for one experimental group through face-to-face/onsite delivery.
  Interventions: Behavioral: The Onsite Nurse-Led Education Programme on IPC
- The Online Nurse-Led Education Programme on IPC (Experimental): The researcher will conduct the Nurse-Led Education Programme on IPC for another experimental group through online platform delivery.
  Interventions: Behavioral: The Online Nurse-Led Education Programme on IPC
- The Control Group (No Intervention): Participants in the control group will continue their usual practice without receiving any intervention and materials until the post-intervention assessment at six months. After that, the researcher will provide the online or onsite programmes and distribute all materials.

INTERVENTIONS:
Behavioral: The Onsite Nurse-Led Education Programme on IPC — The programme was designed to enhance CCWs' IPC knowledge and attitudes through lectures, interactive discussions, information sharing, and Q&A sessions. It also aims to improve their IPC practices and self-efficacy through demonstrations, role-playing exercises, and a work assignment focused on IPC self-monitoring.
  The programme includes five educational sessions totalling 12 hours, along with one session for work assignment on daily self-monitoring of IPC practices over five days. The educational sessions cover the following topics:
  1. General concepts of infectious diseases
  2. Vaccination
  3. Standard precautions: The use of personal protective equipment, environmental cleaning and disinfection, handling food and feeding, and waste management
  4. Standard precautions: Hand hygiene
  5. Common infectious diseases in DCCs and management.
  Arms: The Onsite Nurse-Led Education Programme on IPC
Behavioral: The Online Nurse-Led Education Programme on IPC — The online version of the nurse-led education programme was conducted using an online meeting platform. It includes the same content, learning activities, and materials as the onsite delivery programme, except for the practice stations, which cannot be provided to participants in the online delivery. Additionally, all documents will be available for download via the online platform.
  Arms: The Online Nurse-Led Education Programme on IPC

SUMMARY:
The goal of this clinical trial is to evaluate the effects of nurse-led education programmes on childcare workers (CCWs) in improving infection prevention and control (IPC) practices in daycare centres. The main questions it aims to answer are:

1. Is there an increase in IPC knowledge, attitudes, practices, and self-efficacy, as well as hand hygiene intention and compliance of CCWs after receiving the online or onsite IPC nurse-led education programme?
2. Do CCWs who receive the online programme exhibit higher IPC knowledge, attitudes, practices, and self-efficacy, as well as hand hygiene intention and compliance compared to those who do not receive any programme?
3. Do CCWs who receive the onsite programme exhibit higher IPC knowledge, attitudes, practices, and self-efficacy, as well as hand hygiene intention and compliance compared to those who do not receive any programme?
4. Is there a difference in IPC knowledge, attitudes, practices, and self-efficacy, as well as hand hygiene intention and compliance between CCWs who receive the online programme and those who receive the onsite programme?

DETAILED DESCRIPTION:
Despite the crucial role of infection prevention and control (IPC) in daycare centers (DCCs), research reveals significant gaps. Based on the systematic review of the IPC programmes among childcare workers (CCWs), most studies focus mainly on hand hygiene, neglecting other IPC components like environmental cleaning, waste management, vaccination, and triage of infectious disease patients. Research on the role of nurses in developing and implementing these programmes is also limited. Existing studies often emphasize outcomes related to children and parents rather than assessing the impact on CCWs. Only two studies used a cluster randomized controlled trial (RCT) design, essential for evaluating group interventions.

Additionally, the emergence of online, on-demand, and hybrid learning methods highlights a gap in IPC training, with limited exploration of online learning for IPC education. Comprehensive IPC programmes for CCWs, incorporating various IPC components, clearly defined roles for nurses, and modern educational methods, are urgently needed. These programmes should be rigorously evaluated using cluster RCT designs to provide robust evidence of their effectiveness. Therefore, this clinical trial is aimed to evaluate the effects of nurse-led education programmes on IPC knowledge, attitudes, and practices, as well as hand hygiene intention and compliance among CCWs in daycare centres in Bangkok, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Registered DCCs in Bangkok, as listed in the Bangkok Metropolis Administrative information.
* At least two or more CCWs work in DCC at the time of recruitment.
* Participants aged 18 years or over.
* Participants had been employed for at least three months at registered DCCs in Bangkok at the time of recruitment.
* Participants provided care for children 0-5 years of age.
* Participants could read and speak Thai language.

Exclusion Criteria:

* Participants are attending any IPC training at the time of recruitment.
* Participants are planning to attend another IPC training within six months after the time of recruitment.
* Participants have completed another IPC training programme within the six months prior to the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Infection prevention and control knowledge | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was adapted from an existing validated tool, the knowledge of preventive behaviors for communicable diseases questionnaire. It was developed based on the Disease-Free Child Care Centers Policy from the Department of Disease Control, Thailand Ministry of Public Health, to assess Thai CCWs. The original questionnaire consists of 15 dichotomous questions. The item objective congruence (IOC) was evaluated by five experts, resulting in a score of 0.744, and internal consistency was assessed with a KR-20 of 0.73 (n = 30).
  In this study, the researchers added five questions regarding the knowledge of using personal protective equipment, handling food and feeding, and managing waste. Therefore, the final version of this questionnaire consists of 20 dichotomous questions. The total score will be calculated by summing the correct responses, with higher scores indicating greater levels of IPC knowledge.
Infection prevention and control attitudes | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was adapted from an existing validated tool, the attitudes of preventive behaviors for communicable disease questionnaire. It was developed based on the Disease-Free Child Care Centers Policy from the Department of Disease Control, Thailand Ministry of Public Health, to assess Thai CCWs. The original questionnaire consists of 15 items with five-point Likert scales. The IOC was evaluated by five experts, resulting in a score of 0.744, and internal consistency was assessed with a Cronbach's α of 0.71 (n = 30).
  In this study, the researchers removed questions that were outside the conceptual definition and added questions regarding beliefs, perceptions, and feelings about the importance and necessity of IPC measures. The final version of this questionnaire still consists of 15 items, including both positive and negative statements, with five-point Likert scales. The total score will be calculated, with higher scores indicating more positive attitudes toward IPC.
Infection prevention and control practices | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was adapted from an existing validated tool, the preventive behaviours for communicable disease questionnaire. It was developed based on the Disease-Free Child Care Centers Policy from the Department of Disease Control, Thailand Ministry of Public Health, to assess Thai CCWs. The original questionnaire consists of 15 items with five-point Likert scales. The IOC was evaluated by five experts, resulting in a score of 0.744, and internal consistency was assessed with a Cronbach's α of 0.71 (n = 30).
  In this study, the researchers added five questions regarding practice of vaccination monitoring, the use of personal protective equipment (PPE), handling food and feeding, and waste management. Therefore, the final version of this questionnaire consists of 20 items with five-point Likert scales. The total score will be calculated, with higher scores indicating higher levels of IPC practices.
Infection prevention and control self-efficacy | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was translated and adapted from and existing validated tool, the infectious diseases prevention self-efficacy questionnaire. It was originally used to assess self-efficacy in infectious disease prevention among Korean daycare center administrators. The questionnaire consists of 15 items with five-point Likert scales. The original tool demonstrated internal consistency with a Cronbach's α of 0.91 (n = 172).
  In this study, the original questionnaire was translated from English to Thai by following the WHO guidelines for the process of translation and adaptation of instruments. Additionally, the researchers removed questions that were outside the conceptual definition and added items regarding confidence in the use of PPE, handling food and feeding, and waste management. The final version of the questionnaire still consists of 15 items with five-point Likert scales. The total score will be calculated, with higher scores indicating higher levels of IPC self-efficacy.

SECONDARY OUTCOMES:
Hand hygiene intention | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was translated from an existing validated tool, the hand hygiene intention questionnaire. It was originally developed based on the Theory of Planned Behavior and identified through focus group discussions with caregivers and managers of DCCs to assess hand hygiene intention among CCWs in the Netherlands. The questionnaire consists of 2 items with seven-point Likert scales. The internal consistency was measured with a Cronbach's α of 0.90 (n = 350). The total score will be calculated, with higher scores indicating greater levels of hand hygiene intention.
Hand hygiene compliance | From enrollment to the end of the programme at immediatly, 1 month, 3 months, and 6 months
  This questionnaire was translated and adapted from and existing validated tool, the hand hygiene compliance questionnaire. It was originally developed and commonly used in hand hygiene surveys of caregivers in Netherlands DCCs. The questionnaire consists of 18 items with eleven-point rating scales. It was later used to assess hand hygiene compliance among Chinese kindergarten teachers, reporting an internal consistency with a Cronbach's α of 0.83 (n = 95).

CONTACTS AND LOCATIONS:
Overall Officials: Chakkrich Pidjadee, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Suan Sunandha Rajabhat University, Bangkok, Dusit, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shin J, You SY. The mediating effect of self-efficacy in the relationship between communication skills and practices of preventing infectious diseases among daycare center teachers in South Korea. Child Health Nurs Res. 2021 Jan;27(1):56-64. doi: 10.4094/chnr.2021.27.1.56. Epub 2021 Jan 31. PMID 35004497
- [Background] Zomer TP, Erasmus V, van Empelen P, Looman C, van Beeck EF, Tjon-A-Tsien A, Richardus JH, Voeten HA. Sociocognitive determinants of observed and self-reported compliance to hand hygiene guidelines in child day care centers. Am J Infect Control. 2013 Oct;41(10):862-7. doi: 10.1016/j.ajic.2012.11.023. Epub 2013 Mar 17. PMID 23510663
- [Background] Zomer TP, Erasmus V, Looman CW, VAN Beeck EF, Tjon-A-Tsien A, Richardus JH, Voeten HA. Improving hand hygiene compliance in child daycare centres: a randomized controlled trial. Epidemiol Infect. 2016 Sep;144(12):2552-60. doi: 10.1017/S0950268816000911. Epub 2016 May 19. PMID 27193613
- [Background] Rosen L, Zucker D, Brody D, Engelhard D, Manor O. The effect of a handwashing intervention on preschool educator beliefs, attitudes, knowledge and self-efficacy. Health Educ Res. 2009 Aug;24(4):686-98. doi: 10.1093/her/cyp004. Epub 2009 Mar 24. PMID 19318523
- [Background] Mendes PME, de Jesus Mateus LV, Costa P. Does a Playful Intervention Promote Hand Hygiene? Compliance and Educator's Beliefs about Hand Hygiene at a Daycare Center. J Pediatr Nurs. 2020 Mar-Apr;51:e64-e68. doi: 10.1016/j.pedn.2019.08.017. Epub 2019 Sep 3. PMID 31492509
- [Background] Pidjadee C, Soh KL, Attharos T, Soh KG. The effect of infection prevention and control programme for childcare workers in daycare centres: A systematic review. J Pediatr Nurs. 2024 Nov-Dec;79:116-125. doi: 10.1016/j.pedn.2024.09.002. Epub 2024 Sep 9. PMID 39255691
- See also: Related Info — https://he02.tci-thaijo.org/index.php/PRIJNR/article/view/256513
- See also: Related Info — https://iris.who.int/handle/10665/376810